CLINICAL TRIAL: NCT06568146
Title: A Single Group Study to Evaluate the Effects of a Multivitamin on a Range of Health and Wellbeing Outcomes.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Love Wellness (Industry)
Collaborators: Citruslabs (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 20432
Record Dates: First submitted 2024-07-11; First posted 2024-08-23 (Actual); Last update posted 2024-10-29 (Actual); Status verified 2024-10

CONDITIONS: Health and Wellbeing
Keywords: Multivitamin; Cognitive Function; Iron; Vitamin D; Vitamin B12; Insulin
MeSH Terms: conditions — Insulin Resistance

STUDY DESIGN:
Intervention Model Description: This is a hybrid single-group clinical trial designed to evaluate the effects of a multivitamin on a range of health and wellbeing outcomes over a 12-week period.
Masking Description: This is an open-label study where no masking will be implemented.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Multivitamin Supplement Group (Experimental): Participants in this arm will take 2 capsules of the multivitamin supplement daily with the first meal of the day in the morning.
  Interventions: Dietary Supplement: Multivitamin Supplement

INTERVENTIONS:
Dietary Supplement: Multivitamin Supplement — : Participants will take 2 capsules of the multivitamin supplement daily with the first meal of the day in the morning.
  Other Names: Daily Love Multivitamin

SUMMARY:
This is a hybrid single-group clinical trial that will last 12 weeks. Participants will take 2 capsules daily with the first meal of the day in the morning. Participants will undertake blood tests at Baseline and Week 12. Study-specific questionnaires will be completed at Baseline, Week 4, Week 8, and Week 12. Cognitive Battery Testing will take place at Baseline, Week 4, Week 8, and Week 12.

ELIGIBILITY:
Inclusion Criteria:

* Female at birth.
* Aged 18+.
* Interested in supporting their health and wellbeing.
* Not planning to introduce or change prescription medications, vitamins, minerals, or supplements one month prior to and during the study.
* Generally healthy with no uncontrolled chronic conditions.

Exclusion Criteria:

* Recent surgeries or invasive treatments.
* Introduction of new health-related products in the last 12 weeks.
* Allergies to product ingredients or use of Epi-Pen.
* Chronic health conditions affecting participation.
* Endocrine or glucose-related disorders, including diabetes.
* Hematological disorders, including anemia.
* Pregnant, breastfeeding, or planning to conceive.
* History of substance abuse or recent smoking.
* Unwillingness to follow the study protocol.
* Participation in other clinical trials.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2024-05-23 (Actual); Primary Completion 2024-10-23 (Actual); Study Completion 2024-10-23 (Actual)

PRIMARY OUTCOMES:
Changes in Blood Levels of Vitamin B12 | Baseline and Week 12
  This outcome measure will assess the effect of the multivitamin supplement on serum levels of Vitamin B12.
Changes in Blood Levels of Insulin | Baseline and Week 12
  This outcome measure will assess the effect of the multivitamin supplement on serum levels of Insulin.
Changes in Blood Levels of Vitamin D | Baseline and Week 12
  This outcome measure will assess the effect of the multivitamin supplement on serum levels of Vitamin D.
Changes in Blood Levels of Iron | Baseline and Week 12
  This outcome measure will assess the effect of the multivitamin supplement on serum levels of Iron.

SECONDARY OUTCOMES:
Participants' Perceptions of Health and Wellbeing | Baseline, Week 4, Week 8, and Week 12
  Evaluation of participants' perceptions via a questionnaire exploring the convenience and efficacy of the multivitamin supplement in supporting overall health and wellbeing.

CONTACTS AND LOCATIONS:
Locations (1):
- Citruslabs, Santa Monica, California, United States

IPD SHARING:
Plan to Share IPD: No